CLINICAL TRIAL: NCT01146730
Title: At Work and Coping - Effect Evaluation of Center for Workcoping for Patients With Anxiety and Depression
Brief Title: At Work and Coping - Effect Study of Workcoping for Patients With Anxiety and Depression
Acronym: AWaC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NORCE Norwegian Research Centre AS (Other)
Collaborators: Norwegian Labour and Welfare Administration (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Workcoping2010
Record Dates: First submitted 2010-06-01; First posted 2010-06-17 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Anxiety; Depression
Keywords: Anxiety; Depression; Vocational Rehabilitation; Common Mental Disorders; Mental Health Problems; Work Related Therapy
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Myo-Inositol-1-Phosphate Synthase; Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Workcoping and IPS (Experimental): CBT based counseling and supported employment
  Interventions: Behavioral: Workcoping and IPS
- Ordinary care by GP or NAV (Active Comparator): Ordinary care by GP or The Norwegian Labour and Welfare Administration (NAV)
  Interventions: Behavioral: Ordinary care by GP or NAV

INTERVENTIONS:
Behavioral: Workcoping and IPS — Maximum 15 sessions of CBT-based counseling with workcoping as primary focus in addition to work support according to the IPS-model (individual placement and support)
  Other Names: Cognitive behavior therapy; Cognitive Counseling
  Arms: Workcoping and IPS
Behavioral: Ordinary care by GP or NAV — Ordinary care by the participants physician or the local Labour and Welfare Administration
  Other Names: Treatment as usual
  Arms: Ordinary care by GP or NAV

SUMMARY:
Mental disorders, mainly various anxiety and depressive disorders, are an increasing reason for sick leave and disability pension. Cognitive behaviour therapy (CBT) has been shown to have an effect on anxiety and depression, but the investigators know little about this in relation to employment. Close follow-up in ordinary employment increase employment participation for serious mental illness, but this is not yet investigated to the same degree for lighter mental disorders.

Center for Work-Coping (No: "Senter for Jobbmestring" - SJM) combines Cognitive behaviour therapy (CBT) and individual placement and support (IPS) and facilitation of work for people with anxiety and depression who are in danger of falling out of work.

The purpose of this project is to evaluate the effectiveness of the model in SJM. The effect will be evaluated through a randomized controlled trial (RCT) in which participants will be randomized to SJM or regular follow-up by The Norwegian Labour and Welfare Administration (NAV) or by their regular general practitioners (GP) and self-help resources. The main outcome measures are work participation with changes in mental health as a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Problems coping with work due to psychological illness (anxiety and depression)
* Reasonable closeness to work (possible to return within a year)

Exclusion Criteria:

* Other reasons as primary cause of work problems
* Serous psychiatric disorders
* Suicide risk
* Pregnancy
* Ongoing psychological treatment (therapy)
* Ongoing substance abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1202 (Actual)
Dates: Start 2010-06; Primary Completion 2016-03 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Sick leave data | One year
  The primary outcome of the study is return to work measured through register data.

SECONDARY OUTCOMES:
Psychopathology | 6 and 12 months of follow up
  Secondary outcomes are reductions in psychopathology measured through validated questionnaires (e.g. HADS).

CONTACTS AND LOCATIONS:
Overall Officials: Silje E Reme, PhD, Principal Investigator — NORCE Norwegian Research Centre AS
Locations (1):
- Uni Reserach, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lovvik C, Overland S, Hysing M, Broadbent E, Reme SE. Association between illness perceptions and return-to-work expectations in workers with common mental health symptoms. J Occup Rehabil. 2014 Mar;24(1):160-70. doi: 10.1007/s10926-013-9439-8. PMID 23595310
- [Result] Lovvik C, Shaw W, Overland S, Reme SE. Expectations and illness perceptions as predictors of benefit recipiency among workers with common mental disorders: secondary analysis from a randomised controlled trial. BMJ Open. 2014 Mar 3;4(3):e004321. doi: 10.1136/bmjopen-2013-004321. PMID 24589824
- [Result] Reme SE, Grasdal AL, Lovvik C, Lie SA, Overland S. Work-focused cognitive-behavioural therapy and individual job support to increase work participation in common mental disorders: a randomised controlled multicentre trial. Occup Environ Med. 2015 Oct;72(10):745-52. doi: 10.1136/oemed-2014-102700. Epub 2015 Aug 6. PMID 26251065
- [Result] Overland S, Grasdal A, Reme SE. Trial participant representativeness compared to ordinary service users in a work rehabilitation setting. Contemp Clin Trials Commun. 2015 Dec 17;2:12-15. doi: 10.1016/j.conctc.2015.12.005. eCollection 2016 Apr 15. PMID 29736442
- [Result] Olsen IB, Overland S, Reme SE, Lovvik C. Exploring Work-Related Causal Attributions of Common Mental Disorders. J Occup Rehabil. 2015 Sep;25(3):493-505. doi: 10.1007/s10926-014-9556-z. PMID 25451074
- [Derived] Overland S, Grasdal AL, Reme SE. Long-term effects on income and sickness benefits after work-focused cognitive-behavioural therapy and individual job support: a pragmatic, multicentre, randomised controlled trial. Occup Environ Med. 2018 Oct;75(10):703-708. doi: 10.1136/oemed-2018-105137. Epub 2018 Jul 21. PMID 30032103
- See also: Study website — http://uni.no/nb/uni-helse/stress-helse-og-rehabilitering/effektevaluering-av-senter-for-jobbmestring/